CLINICAL TRIAL: NCT04228289
Title: Enhancing Prolonged Exposure Therapy for PTSD With Oxytocin
Brief Title: Oxytocin to Treat PTSD
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Collaborators: San Francisco VA Health Care System (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MHBB-001-19S
Record Dates: First submitted 2019-12-30; First posted 2020-01-14 (Actual); Last update posted 2025-09-11 (Actual); Status verified 2025-09

CONDITIONS: PTSD
Keywords: PTSD; Veterans; Oxytocin; Mental Health; Psychophysiology
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Psychological Well-Being | interventions — Oxytocin; Sodium Chloride

STUDY DESIGN:
Intervention Model Description: Participants will be randomized in a 1:1 manner to one of two drug conditions
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Oxytocin (Experimental): 40 IU intranasal oxytocin
  Interventions: Drug: Oxytocin
- Placebo (Placebo Comparator): intranasal saline spray
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Oxytocin — 40 IU intranasal spray
  Other Names: Pitocin
  Arms: Oxytocin
Other: Placebo — matching intranasal spray
  Other Names: Saline
  Arms: Placebo

SUMMARY:
Posttraumatic stress disorder (PTSD) is a chronic, debilitating condition that disproportionately affects Veterans. Prolonged Exposure (PE) therapy is a "gold standard" treatment for PTSD. However, approximately one-third of Veterans fail to receive an adequate dose of treatment because they prematurely drop out of PE therapy. There is also room to improve PE treatment outcomes. Consistent with the VA Office of Research and Development initiative to develop effective treatments for PTSD, the proposed randomized clinical trial will examine the ability of oxytocin (as compared with placebo) combined with PE to reduce PTSD symptom severity, improve the rate of PTSD symptom reduction, and to enhance PE treatment retention and adherence. This two-site study will leverage the investments made in the nationwide rollout off PE therapy and has the potential to significantly improve mental health care among Veterans, advance the science in this area, and identify mechanisms underlying positive PTSD treatment response. Participants may choose to complete this research study via home-based telemedicine (HBT) care (i.e. service delivery to patients in their homes using consumer friendly, video-conferencing technology). HBT sessions will be delivered via standard desk, laptop computer, tablet, or smartphone using VA approved applications. All procedures that take place via telemedicine will be performed and completed as though they were in-person/in-office

DETAILED DESCRIPTION:
Posttraumatic stress disorder (PTSD) is the most highly prevalent mental health disorder among U.S. military Veterans. PTSD is a chronic disorder that is associated with significant morbidity, mortality, disability, and costly health care expenditures. The clinical impairment associated with PTSD among Veterans is severe and associated with comorbid depression, suicidality, substance abuse, physical health problems, interpersonal violence, and neuropsychiatric impairment. Despite these pervasive health consequences, the current treatment services offered to Veterans do not adequately address PTSD. Several promising psychosocial interventions, including Prolonged Exposure (PE) therapy, have been developed for the treatment of PTSD. Although PE is one of the most widely used evidence-based treatments for PTSD, there is substantial room for improvement in outcomes and retention rates. For example, approximately one-third of patients dropout of PE treatment prematurely, and the highest dropout rates occur among Veterans. Consistent with the VA Office of Research and Development initiative to develop effective treatments for PTSD, identifying pharmacotherapies to enhance PTSD treatment retention and outcomes is critical. Accumulating data from the investigators' group and others suggests that oxytocin is a promising candidate to achieve this goal. Oxytocin is known to promote prosocial behaviors associated with successful psychosocial treatment outcomes (e.g., trust, safety, social cognition) and has demonstrated positive effects on extinction learning in animal and human stress models. Furthermore, recent neuroimaging studies show that oxytocin has the ability to ameliorate dysregulation of the corticolimbic brain circuitry, which is a central component of the pathophysiology and maintenance of PTSD. In the only study to date examining the feasibility, acceptability, and preliminary efficacy of augmenting PE with oxytocin, the investigators' group found that participants randomized to the oxytocin condition demonstrated lower PTSD and depression symptoms during PE, and had higher working alliance scores compared to participants randomized to the placebo condition. Therefore, the primary objective of the proposed two-site Phase II study is to examine the ability of oxytocin (vs. placebo) combined with PE therapy to (1) reduce PTSD symptom severity, (2) improve rate of PTSD symptom improvement, and (3) improve PE adherence and retention rates. To accomplish these objectives, the investigators will employ a randomized, double-blind, placebo-controlled trial and use standardized, repeated dependent measures of change at five time points (baseline, mid-treatment, end of treatment, and 3 and 6 month follow-up). The proposed study directly addresses the mission of the Veterans Health Administration Blueprint for Excellence in that it seeks to advance personalized and proactive mental health care opportunities for Veterans. Findings from this study will provide critical new information regarding the efficacy of oxytocin to augment psychosocial treatment for PTSD, as well as information regarding the neurobiological mechanisms underlying PTSD and positive treatment response. Participants may choose to complete this research study via home-based telemedicine (HBT) care (i.e. service delivery to patients in their homes using consumer friendly, video-conferencing technology). HBT sessions will be delivered via standard desk, laptop computer, tablet, or smartphone using VA approved applications. All procedures that take place via telemedicine will be performed and completed as though they were in-person/in-office

ELIGIBILITY:
Inclusion Criteria:

* Veteran
* Any race or ethnicity
* Able to provide informed consent and function at an intellectual level sufficient to allow accurate completion of the assessment instruments (> 26 on the Mini Mental Status Exam)
* Meet DSM-5 diagnostic criteria for current (i.e., past 6 months) PTSD (assessed via the CAPS-5)

  * participants may also meet criteria for a mood disorder (except bipolar affective disorder, see Exclusion Criteria)
  * anxiety disorders (e.g. panic disorder, agoraphobia, social phobia, generalized anxiety disorder, or obsessive compulsive disorder)
* Participants taking psychotropic medications will be required to be maintained on a stable dose for at least four weeks before study initiation

Exclusion Criteria:

* Meeting DSM-5 criteria for a history of or current psychotic or bipolar affective disorders, or with current suicidal or homicidal ideation and intent

  * those participants will be referred clinically
* Participants who present a serious suicide risk or are likely to require hospitalization during the study
* Participants on maintenance anxiolytic, antidepressant, or mood stabilizing medications, which have been initiated during the past 4 weeks
* Pregnancy or breastfeeding for women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 185 (Actual)
Dates: Start 2020-11-16 (Actual); Primary Completion 2025-02-28 (Actual); Study Completion 2025-08-31 (Actual)

PRIMARY OUTCOMES:
PTSD symptom severity as measured by the Clinician-Administered PTSD Scale (CAPS-5) | End of Treatment (10 weeks)
  Total CAPS-5 Scores range from 0-80. Higher scores indicate greater symptom severity.
PTSD Symptom Severity as measured by the PTSD Checklist (PCL-5) | End of Treatment (10 weeks)
  Total PCL-5 Scores range from 17-85. Higher scores indicate greater symptom severity.

SECONDARY OUTCOMES:
Number of sessions attended | End of Treatment (10 weeks)
  Total number of sessions attended during the treatment phase
Number of homework assignments completed | End of Treatment (10 weeks)
  Total number and proportion of completed homework assignments during treatment phase

CONTACTS AND LOCATIONS:
Overall Officials: Julianne Christina Flanagan, PhD, Principal Investigator — Ralph H. Johnson VA Medical Center, Charleston, SC
Locations (2):
- United States (2):
  - San Francisco VA Medical Center, San Francisco, CA, San Francisco, California
  - Ralph H. Johnson VA Medical Center, Charleston, SC, Charleston, South Carolina

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Flanagan JC, Mitchell JM, Baker NL, Woolley J, Wangelin B, Back SE, McQuaid JR, Neylan TC, Wolfe WR, Brady KT. Enhancing prolonged exposure therapy for PTSD among veterans with oxytocin: Design of a multisite randomized controlled trial. Contemp Clin Trials. 2020 Aug;95:106074. doi: 10.1016/j.cct.2020.106074. Epub 2020 Jun 16. PMID 32561468

DOCUMENTS (1):
  • Informed Consent Form (2024-09-04): https://cdn.clinicaltrials.gov/large-docs/89/NCT04228289/ICF_000.pdf